CLINICAL TRIAL: NCT00985413
Title: An Observational Study to Assess the Natural History Including Growth and Hearing in Patients With Cockayne Syndrome
Brief Title: Observational Study to Assess Natural History in Cockayne Syndrome Patients
Status: Terminated | Type: Observational
Why Stopped: The company DNage is in receivership and no longer functional
Sponsor: DNage B.V. (Industry)
Responsible Party: Dr. E. Neilan, Principal Investigator, Children's Hospital Boston
Other Study IDs: MP1003-01; NCT01230333 (obsolete NCT alias)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Cockayne Syndrome
Keywords: Cockayne Syndrome; pediatrics; growth; hearing; Ageing
MeSH Terms: conditions — Cockayne Syndrome

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — whole blood, plasma, serum, white blood cells, urine, tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an Observational Study of children under the age of 11 diagnosed with Cockayne Syndrome to assess the natural progression of Cockayne Syndrome disease, with special attention to hearing and physical changes in length or height, weight, head circumference, and arm span during standard treatment.

The primary analytical objective is to determine the rate of linear growth over a 6-month period in children < 2 years of age and over a 12-month period in children ≥ 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with a documented diagnosis of CS, as suggested by clinical features and possible confirmation by genetic consultation and analysis
* Age of participation:

  * At least 12 months of age at the time of signing Informed Consent/Assent
  * Female patient's age will not be greater than 10 years of age at the time of signing Informed Consent/Assent
  * Male patient's age will not be greater than 11 years of age at the time of signing Informed Consent/Assent

Exclusion Criteria:

* Severe contractures or physical deformities that in the opinion of the investigator would prevent accurate measurement of height, length and ulna length
* Patients that have taken growth hormone or growth hormone related medications within 12 months prior to the date of Informed Consent/Assent
* Known history of inborn error of hyperprolinemia (Type I or Type II)
* Clinical features present at the time of initial screening that are associated with the terminal phases of the natural progression of CS suggesting safe travel and completion of the study and its assessments to be unlikely as judged by the Investigator, including any of the following:

  * Continuous or intermittent dependence on supplemental oxygen at home during the prior six months
  * Two or more hospitalizations for pneumonia during the prior 12 months;
  * A documented net weight loss of at least 10%, which has not been recovered and which includes a significant net weight loss (beyond the estimated error of the measurement) over the most recent 6 months, despite intensive nutritional support including the use of gastrostomy tube feedings
* Presence of scoliosis with a Cobb's angle of 30º or greater

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients up to 10 years of age for females and up to 11 years of age for males who have received a diagnosis of Cockayne Syndrome
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the rate of linear growth over a 6-month period in children < 2 years of age and over a 12-month period in children ≥ 2 years of age. | 6 -12 months

SECONDARY OUTCOMES:
Hearing Test Results tabulated and with the severity/deficits to be correlated with patient age, height velocity, and Pediatric Evaluation of Disabilities Inventory (PEDI)Score | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: E. G. Neilan, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (4):
- United States (2):
  - Harvard medical School, Children's Hospital Boston, Division of Genetics & Metabolism, Boston, Massachusetts
  - New York University Medical Center, New York, New York
- Hopitaux Universitaires de Strasbourg, Service de Pédiatrie 1, Strasbourg, Cedex, France
- St. Mary's Hospital, Genetic Medicine, 6th Floor, Oxford Road, Manchester, United Kingdom